CLINICAL TRIAL: NCT00692705
Title: Open Label Positron Emission Tomography (PET) Study With [11C]AZD2995 and [11C]AZD2184, Candidate PET Ligands for β Amyloid, to Determine and Compare in Vivo Brain Uptake and Distribution in Healthy Volunteers and Patients With Alzheimer's Disease
Brief Title: Positron Emission Tomography (PET) Study With [11C]AZD2995 and [11C]AZD2184, Candidate PET Ligands for β Amyloid
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Märta Segerdahl, Medical Science Director, AstraZeneca, Research and Development, Sweden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D0180C00018; Eudract No. 2007-004842-33
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Alzheimer´s Disease
Keywords: Alzheimer´s Disease; amyloid deposits; Positron Emission Tomography; phase I
MeSH Terms: conditions — Plaque, Amyloid | interventions — AZD2995

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Alzheimer's Disease (AD) patients
  Interventions: Drug: Radioligand (11C)AZD2995; Drug: Radioligand (11C)AZD2184
- 2 (Other): Healthy volunteers
  Interventions: Drug: Radioligand (11C)AZD2995; Drug: Radioligand (11C)AZD2184

INTERVENTIONS:
Drug: Radioligand (11C)AZD2995 — Single dose of i.v solution. 1-2 times for AD patients. Once for healthy volunteers.
Drug: Radioligand (11C)AZD2184 — Single dose of i.v solution. Once for AD patients respective healthy volunteers.

SUMMARY:
The study is carried out in order to investigate if [11C]AZD2995, compared to [11C]AZD2184, is a more suitable PET ligand for in vivo imaging of β amyloid depositions in the human brain. In the study the two PET ligands will be examined in both healthy volunteers and patients with Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer´s Disease patients - 50-85 years- mild to moderate AD, clinical progression of AD over 12 months.
* Healthy male volunteers: - Age 20-50 years, Body Mass Index: 18-30 kg/m2.
* Clinically normal physical findings including normal blood pressure and pulse rate.

Exclusion Criteria:

* Alzheimer´s Disease patients:
* significant cerebrovascular disease or depression, central nervous system infarct or infection or lesions
* clinically significant illness within 2 weeks before the study start.
* administration of any investigational product with effect on brain beta amyloid levels within 3 months prior to study and/or participation in a PET investigation other than study D0180C00011 as part of a scientific study during the past 12 months,.
* Healthy volunteers; - clinically significant illness within 2 weeks before the study start, history of psychiatric or somatic disease/condition that may interfere.- first degree relative with dementia. Obvious deterioration of memory functions.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography using the radioligand (11C)AZD2995 or (11C)AZD2184 | Radioligand (11C)AZD2995.1-2 PET examinations for AD patients and 1 PET examination for healthy volunteers. - Radioligand (11C) AZD2184.One PET for AD patients respective healthy volunteers.

SECONDARY OUTCOMES:
To assess safety and tolerability of [11C]AZD2995, [11C]AZD2184 and the study procedures, by assessment of adverse events, vital signs and laboratory variables. | 3-4 visits with tests for the AD patients. 3 visits with tests for the healthy volunteers. All tests are not done at every visit.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Jönhagen, Principal Investigator — Geriatric Clinic, Karolinska University Hospital, Huddinge, Sweden; Ingemar Bylesjö, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Stockholm, Sweden; Emma Gyllenpalm, Study Director — AstraZeneca R&D, Södertälje, Sweden
Locations (1):
- Research Site, Stockholm, Sweden